CLINICAL TRIAL: NCT01968356
Title: Assessment of the Antimicrobial Efficacy of 3M CHG/IPA Preoperative Skin Preparation Against Resident Human Skin Flora on the Abdominal and Inguinal Regions
Brief Title: In-vivo Efficacy Study of Patient Preoperative Preps
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study discontinued due to data quality issues.
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EM-012759
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Skin Flora Bacterial Reduction Post-product Application
Keywords: surgical skin prep; CHG; IPA
MeSH Terms: interventions — 2-Propanol; Chromogranins; chlorhexidine gluconate; Ethanol; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- 3M CHG/IPA Prep Colorless (Experimental): Applied topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: 3M CHG/IPA Prep Colorless
- 3M CHG/IPA Prep Tint (Experimental): Applied topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: 3M CHG/IPA Prep Tint
- ChloraPrep Hi-Lite Orange (Active Comparator): Applied topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: ChloraPrep
- Normal Saline (Placebo Comparator): Applied topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: 3M CHG/IPA Prep Colorless — Apply topically.
  Other Names: Chlorhexidine glucontate and Isopropyl alcohol; CHG 2% / IPA 70%; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Arms: 3M CHG/IPA Prep Colorless
Drug: 3M CHG/IPA Prep Tint — Apply topically.
  Other Names: Chlorhexidine glucontate and Isopropyl alcohol; CHG 2%/IPA 70%; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Arms: 3M CHG/IPA Prep Tint
Drug: ChloraPrep — Apply topically.
  Other Names: ChloraPrep One-Step; ChloraPrep Patient Preoperative Skin Preparation; 2% CHG/70% IPA; Chlorhexidine glucontate and Isopropyl alcohol; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Arms: ChloraPrep Hi-Lite Orange
Drug: Saline — Apply topically.
  Other Names: 0.9% NaCl; Normal Saline
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to evaluate the antimicrobial efficacy of the 3M CHG/IPA Prep on skin flora of the abdominal and inguinal regions of human subjects.

DETAILED DESCRIPTION:
The primary efficacy is evaluated by demonstration that the product provides a lower bound of the 95% confidence interval of percent responders that is greater than or equal to 70%. On the abdominal sites, a responder is defined as a subject with a 2-log10 per cm2 bacterial reduction at 10 minutes and for whom the skin flora does not return to baseline at 6 hours. On the inguinal sites, a responder is defined as a subject with a 3-log10 per cm2 bacterial reduction at 10 minutes and for whom the skin flora does not return to baseline at 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race
* Subjects in good general health
* Minimum skin flora baseline requirements on abdomen and groin

Exclusion Criteria:

* Any tattoos, scars, breaks in the skin, or any form of dermatitis, or other skin disorders (including acne) on the applicable test areas
* Topical antimicrobial exposure within 14 days prior to screening and treatment days
* Use of systemic or topical antibiotics, steroid medications, or any other products known to affect the normal microbial flora of the skin within 14 days prior to screening and treatment days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R McCormack, BS, Principal Investigator — BioScience Laboratories, Inc.
Locations (1):
- BioScience Laboratories, Inc., Bozeman, Montana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a randomized, paired comparison design where each subject received 2 of the planned treatments, 1 on the left side and one on the right. Each subject provided 2 abdomen test sites, left & right and/or 2 inguen test sites, left & right.
  161 subjects were randomized for the abdomen region & 162 subjects randomized for the inguen region, resulting in 171 subjects providing 646 applications of test products on 2 anatomical regions.
Units Other Than Participants: test sites on skin
Groups:
- 3M CHG/IPA Prep Colorless Abdominal Region; 3M CHG/IPA Prep Colorless Inguinal Region; 3M CHG/IPA Prep Tint Inguinal Region: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 10.5 mL applicator
  3M CHG/IPA Prep Colorless: Apply topically.
- 3M CHG/IPA Prep Tint Abdominal Region: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 10.5 mL applicator
  3M CHG/IPA Prep Tint: Apply topically.
- ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region; ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 10.5 mL applicator
  ChloraPrep CHG/IPA Hi-Lite Orange Tint: Apply topically.
- Normal Saline Abdominal Region; Normal Saline Inguinal Region: 0.9% normal saline with applicator
  Normal Saline: Apply topically.
Period: Overall Study
Arm/Group | 3M CHG/IPA Prep Colorless Abdominal Region | 3M CHG/IPA Prep Tint Abdominal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region | Normal Saline Abdominal Region | 3M CHG/IPA Prep Colorless Inguinal Region | 3M CHG/IPA Prep Tint Inguinal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region | Normal Saline Inguinal Region
Started | 101; 101 test sites on skin | 93; 93 test sites on skin | 96; 96 test sites on skin | 32; 32 test sites on skin | 97; 97 test sites on skin | 99; 99 test sites on skin | 97; 97 test sites on skin | 31; 31 test sites on skin
Completed | 101; 101 test sites on skin | 93; 93 test sites on skin | 96; 96 test sites on skin | 32; 32 test sites on skin | 97; 97 test sites on skin | 99; 99 test sites on skin | 97; 97 test sites on skin | 31; 31 test sites on skin
Not Completed | 0; 0 test sites on skin | 0; 0 test sites on skin | 0; 0 test sites on skin | 0; 0 test sites on skin | 0; 0 test sites on skin | 0; 0 test sites on skin | 0; 0 test sites on skin | 0; 0 test sites on skin

BASELINE CHARACTERISTICS:
Population: Subjects with average screening day baseline counts of > or equal to 3.00 log10 CFU/cm2 bilaterally on the abdominal region and/or > or equal to 5.00 log10 CFU/cm2 bilaterally on the inguinal region were to be included in the efficacy analysis. However, due to early study termination the primary efficacy endpoint analysis was not performed. The 171 subjects who provided 646 test sites on skin for product application on the 2 anatomical regions were included in the safety analyses.
Units Other Than Participants: test sites on skin
Groups:
- Total: Total of all reporting groups
Arm/Group | 3M CHG/IPA Prep Colorless Abdominal Region | 3M CHG/IPA Prep Tint Abdominal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region | Normal Saline Abdominal Region | 3M CHG/IPA Prep Colorless Inguinal Region | 3M CHG/IPA Prep Tint Inguinal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region | Normal Saline Inguinal Region | Total
Number analyzed (Participants) | 101 | 93 | 96 | 32 | 97 | 99 | 97 | 31 | 171
Number analyzed (test sites on skin) | 101 | 93 | 96 | 32 | 97 | 99 | 97 | 31 | 646
Age, Customized [Number; unit: test sites on skin]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 99 | 92 | 94 | 31 | 96 | 96 | 95 | 31 | 634
  >=66 years | 2 | 1 | 2 | 1 | 1 | 3 | 2 | 0 | 12
Sex/Gender, Customized [Number; unit: test sites on skin]
  Sex : Female | 23 | 28 | 27 | 7 | 31 | 22 | 21 | 11 | 170
  Sex : Male | 78 | 65 | 69 | 25 | 66 | 77 | 76 | 20 | 476
Race/Ethnicity, Customized [Number; unit: test sites on skin]
  White | 88 | 86 | 80 | 28 | 84 | 88 | 85 | 25 | 564
  Hispanic/Latino | 2 | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 18
  Black or Africian American | 3 | 0 | 3 | 0 | 1 | 2 | 2 | 1 | 12
  Native Hawaiian or other Pacific Islander | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 8
  American Indian or Alaska Native | 4 | 1 | 4 | 1 | 4 | 4 | 3 | 1 | 22
  Asian | 2 | 1 | 3 | 0 | 3 | 1 | 1 | 1 | 12
  Other | 1 | 2 | 2 | 1 | 1 | 0 | 2 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate
Description: On the abdominal region a responder was a subject with a 2-log10/cm2 bacterial reduction at 10 minutes and for whom the skin flora did not return to baseline at 6 hours.
  On the inguinal region a responder was a subject with a 3-log10/cm2 bacterial reduction at 10 minutes and for whom the skin flora did not return to baseline at 6 hours.
Time Frame: baseline, 10 minute post-product application and 6 hour post-product application
Population: This study was discontinued prematurely due to technical and data quality issues. In agreement with the FDA no efficacy analysis was conducted. Thus, the efficacy objective of the study could not be evaluated.
Arm/Group | 3M CHG/IPA Prep Colorless Abdominal Region | 3M CHG/IPA Prep Tint Abdominal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region | Normal Saline Abdominal Region | 3M CHG/IPA Prep Colorless Inguinal Region | 3M CHG/IPA Prep Tint Inguinal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region | Normal Saline Inguinal Region
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Skin Flora Baseline for Abdominal and Inguinal Regions
Description: Log10/cm2 baseline skin flora for abdominal and inguinal regions
Time Frame: Baseline
Population: as for outcome 1
Arm/Group | 3M CHG/IPA Prep Colorless Abdominal Region | 3M CHG/IPA Prep Tint Abdominal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region | Normal Saline Abdominal Region | 3M CHG/IPA Prep Colorless Inguinal Region | 3M CHG/IPA Prep Tint Inguinal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region | Normal Saline Inguinal Region
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Skin Flora Recovery Post-treatment
Description: Log10/cm2 recovery of skin flora at 10 minutes and 6 hours following application of study treatments for abdominal and inguinal regions
Time Frame: 10 minutes and 6 hours post-treatment
Population: as for outcome 1
Groups:
- 3M CHG/IPA Prep Colorless - Abdominal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 10.5 mL applicator applied topically to the abdominal region for 30 seconds
  3M CHG/IPA Prep Tint: Apply topically.
  ChloraPrep: Apply topically.
  Saline: Apply topically.
- 3M CHG/IPA Prep Tint - Abdominal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 10.5 mL applicator applied topically to the abdominal region for 30 seconds
  3M CHG/IPA Prep Colorless: Apply topically.
  ChloraPrep: Apply topically.
  Saline: Apply topically.
- ChloraPrep Hi-Lite Orange - Abdominal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 10.5 mL applicator applied topically to the abdominal region for 30 seconds
  3M CHG/IPA Prep Colorless: Apply topically.
  3M CHG/IPA Prep Tint: Apply topically.
  Saline: Apply topically.
- Normal Saline - Abdominal: 0.9% normal saline applied topically to the abdominal region with applicator for 30 seconds
  3M CHG/IPA Prep Colorless: Apply topically.
  3M CHG/IPA Prep Tint: Apply topically.
  ChloraPrep: Apply topically.
- 3M CHG/IPA Prep Colorless - Inguinal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 10.5 mL applicator applied topically to the inguinal region for 2 minutes
  3M CHG/IPA Prep Tint: Apply topically.
  ChloraPrep: Apply topically.
  Saline: Apply topically.
- 3M CHG/IPA Prep Tint - Inguinal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 10.5 mL applicator applied topically to the inguinal region for 2 minutes
  3M CHG/IPA Prep Colorless: Apply topically.
  ChloraPrep: Apply topically.
  Saline: Apply topically.
- ChloraPrep Hi-Lite Orange - Inguinal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 10.5 mL applicator applied topically to the inguinal region for 2 minutes
  3M CHG/IPA Prep Colorless: Apply topically.
  3M CHG/IPA Prep Tint: Apply topically.
  Saline: Apply topically.
- Normal Saline - Inguinal: 0.9% normal saline applied topically to the inguinal region with applicator for 2 minutes
  3M CHG/IPA Prep Colorless: Apply topically.
  3M CHG/IPA Prep Tint: Apply topically.
  ChloraPrep: Apply topically.
Arm/Group | 3M CHG/IPA Prep Colorless - Abdominal | 3M CHG/IPA Prep Tint - Abdominal | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Colorless - Inguinal | 3M CHG/IPA Prep Tint - Inguinal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Reduction of Skin Flora Post-treatment
Description: Log10/cm2 reduction of skin flora, relative to Treatment Day baseline log10/cm2, at 10 minutes and 6 hours
Time Frame: Baseline, 10 minutes and 6 hours
Population: as for outcome 1
Arm/Group | 3M CHG/IPA Prep Colorless Abdominal Region | 3M CHG/IPA Prep Tint Abdominal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region | Normal Saline Abdominal Region | 3M CHG/IPA Prep Colorless Inguinal Region | 3M CHG/IPA Prep Tint Inguinal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region | Normal Saline Inguinal Region
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Safety as Assessed by Skin Irritation Scores
Description: Skin irritation rating (0-3) scores for dryness, edema, erythema and rash. 0 = no reaction, 1 = mild, 2 = moderate, 3 = severe. A skin irritation rating of 3 in any category represents significant irritation and qualifies as an adverse event.
Time Frame: Baseline
Population: # of sites treated (met inclusion/exclusion criteria including screening day baseline counts)
Measure: Count of Participants; unit: Participants
Arm/Group | 3M CHG/IPA Prep Colorless Abdominal Region | 3M CHG/IPA Prep Tint Abdominal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region | Normal Saline Abdominal Region | 3M CHG/IPA Prep Colorless Inguinal Region | 3M CHG/IPA Prep Tint Inguinal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region | Normal Saline Inguinal Region
Number analyzed (Participants) | 101 | 93 | 96 | 32 | 97 | 99 | 97 | 31
Participants
  Dryness-No reaction (0) | 101 | 93 | 96 | 32 | 97 | 97 | 96 | 30
  Dryness-Mild (1) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
  Dryness-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dryness-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-No reaction (0) | 101 | 93 | 96 | 32 | 97 | 98 | 96 | 31
  Edema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Edema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema- No reaction (0) | 99 | 90 | 96 | 31 | 97 | 97 | 96 | 30
  Erythema-Mild (1) | 2 | 3 | 0 | 1 | 0 | 2 | 1 | 1
  Erythema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-No Reaction (0) | 101 | 93 | 96 | 32 | 97 | 97 | 96 | 30
  Rash-Mild (1) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
  Rash-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Safety as Assessed by Skin Irritation Scores
Description: as for outcome 5
Time Frame: 10 minutes post-treatment
Population: # of sites treated (met inclusion/exclusion criteria including screening day baseline counts
Measure: Count of Participants; unit: Participants
Arm/Group | 3M CHG/IPA Prep Colorless Abdominal Region | 3M CHG/IPA Prep Tint Abdominal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region | Normal Saline Abdominal Region | 3M CHG/IPA Prep Colorless Inguinal Region | 3M CHG/IPA Prep Tint Inguinal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region | Normal Saline Inguinal Region
Number analyzed (Participants) | 101 | 93 | 96 | 32 | 97 | 99 | 97 | 31
Participants
  Dryness-No Reaction (0) | 101 | 93 | 96 | 32 | 97 | 97 | 96 | 30
  Dryness-Mild (1) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
  Dryness-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dryness-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-No Reaction (0) | 101 | 93 | 96 | 32 | 97 | 98 | 96 | 31
  Edema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Edema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-No Reaction (0) | 98 | 91 | 96 | 31 | 96 | 97 | 96 | 30
  Erythema-Mild (1) | 3 | 2 | 0 | 1 | 1 | 2 | 1 | 1
  Erythema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-No Reaction (0) | 101 | 93 | 96 | 32 | 96 | 97 | 96 | 30
  Rash-Mild (1) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
  Rash-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Safety as Assessed by Skin Irritation Scores
Description: as for outcome 5
Time Frame: 6 hours post-treatment
Population: # sites treated (met inclusion/exclusion criteria including screening day baseline counts)
Measure: Count of Participants; unit: Participants
Arm/Group | 3M CHG/IPA Prep Colorless Abdominal Region | 3M CHG/IPA Prep Tint Abdominal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region | Normal Saline Abdominal Region | 3M CHG/IPA Prep Colorless Inguinal Region | 3M CHG/IPA Prep Tint Inguinal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region | Normal Saline Inguinal Region
Number analyzed (Participants) | 101 | 93 | 96 | 32 | 97 | 99 | 97 | 31
Participants
  Dryness-No Reaction (0) | 101 | 93 | 96 | 32 | 97 | 99 | 97 | 31
  Dryness-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dryness-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dryness-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-No Reaction (0) | 101 | 93 | 96 | 32 | 97 | 99 | 97 | 31
  Edema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-No Reaction (0) | 101 | 93 | 96 | 32 | 97 | 96 | 97 | 30
  Erythema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
  Erythema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-No Reaction (0) | 101 | 93 | 96 | 32 | 97 | 99 | 97 | 31
  Rash-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected on treatment day (1 day), thus all AEs by definition would be treatment-emergent.
Description: On Treatment Day, prior to collection of the baseline, 10-minute, and 6-hour post-prep samples, the skin in each test area will be evaluated for indications of skin irritation (dryness, edema, erythema, rash), based on the Skin Irritation Rating Scale: 0 = no reaction, 1 = mild, 2 = moderate, 3 = severe. A skin irritation rating of 3 in any category represents significant irritation and qualifies as an adverse event.
Arm/Group | 3M CHG/IPA Prep Tint Abdominal Region | 3M CHG/IPA Prep Colorless Abdominal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Abdominal Region | Normal Saline Abdominal Region | 3M CHG/IPA Prep Colorless Inguinal Region | 3M CHG/IPA Prep Tint Inguinal Region | ChloraPrep CHG/IPA Hi-Lite Orange Tint Inguinal Region | Normal Saline Inguinal Region
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/101 | 0/96 | 0/32 | 0/97 | 0/99 | 0/97 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/101 | 0/96 | 0/32 | 0/97 | 0/99 | 0/97 | 0/31
Other Adverse Events (participants affected / at risk) | 0/93 | 0/101 | 0/96 | 0/32 | 0/97 | 0/99 | 0/97 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes